CLINICAL TRIAL: NCT00845806
Title: Neuronal Processing of Diacritics: An fMRI Study
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Mitchell Albert, Director of Advanced MRI Center, UMASS Medical Sch, University of Massachusetts, Worcester
Other Study IDs: Docket # 13127
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Neuronal Processing of Diacritics
Keywords: Diacritics; Neuronal Processing; fMRI; Arabic

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arabic Speakers: All subjects must be male native arabic speakers who can read and speak english.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — All subjects will be asked to lay in an MRI for about an hour while reading Arabic diacritic characters
  Other Names: Arabic; Diacritic; fMRI

SUMMARY:
The purpose of this study is to determine brain function in reading arabic diacritics.

DETAILED DESCRIPTION:
fMRI is a well established imaging technique that allows investigators to see regional brain function based off of actions like reading, speaking, playing music, etc. Even the type of language and format of that language can change the area of the brain that is active while performing that action. This study is meant to see the areas of the brain that become active both prior to and during the process of reading diacritic markings in arabic.

ELIGIBILITY:
Inclusion Criteria

Adult patients may be enrolled in this study if they meet the following inclusion criteria:

* Are male and are 18 years or older, inclusive;
* Consent from the patient
* First language is Arabic
* Must be able to speak and read English
* Right handed
* The subject must pass a dyslexia screen test (Attached to consent form).

Exclusion Criteria

Adult patients will be excluded from this study if they do not fulfill the inclusion criteria, or if any of the following conditions have been met:

* Have any contraindications to an MR exam such as a pace-maker, metallic cardiac valves, magnetic material (i.e., surgical clips) implanted electronic infusion pumps or any other conditions that would preclude proximity to a strong magnetic field;
* Are undergoing the MR exam in an emergency situation
* People with psychiatric disorders will be excluded from the study.
* Are claustrophobic and can not tolerate the imaging.
* People with neurological diseases
* Are on any medications for psychiatric, neurological, or chronic pain problems.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects will be male native arabic speakers that can read and write english. All will be healthy with no history of neurological or psychiatric disorders.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Observe regional brain function from reading Arabic diacritics | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Albert, Ph.D., Principal Investigator — UMASS Medical School
Locations (1):
- UMASS Medical School Advanced MRI Center, Worcester, Massachusetts, United States